CLINICAL TRIAL: NCT00167908
Title: Pilot Study to Test Whether Amifostine Can Further Protect Salivary Function in Head and Neck Cancer Patients Treated With IMRT
Brief Title: Study of Amifostine and IMRT for Protecting Salivary Glands in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Wade Thorstad, MD, Washington University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETH018-01D; HSC 00-0885
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Amifostine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Ethyol (drug)

SUMMARY:
The purpose of this study is to determine whether Amifostine provides additional protection of salivary gland function over that achieved with IMRT alone.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed squamous cell cancer of the head and neck
* Eligible sites: oral cavity, oropharynx, hypopharynx, larynx.
* Patients requiring postoperative IMRT.
* KPS > 70%.
* Patient has signed specific protocol consent prior to registration.
* Calcium test within normal limits.
* No previous malignancy except for non-melanoma skin cancer or cancer not of head and neck and controlled for at least 5 years.
* Labs completed with 30 days of registration (CBC & platelet, Ca++, Alk phos, SGOT, Bili, albumin) CXR and CT simulation.
* Liver CT if alk phos, SGOT, or bili elevated.
* Bone scan if elevated alk phos

Exclusion Criteria:

* Metastatic disease.
* Patient using Salagen or concurrent chemotherapy.
* Previous XRT for head and neck tumors.
* Active untreated infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2001-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Salivary function at 6 months and yearly compared to pre-treatment salivary function

SECONDARY OUTCOMES:
Local and regional tumor control

CONTACTS AND LOCATIONS:
Overall Officials: Wade Thorstad, M.D., Principal Investigator — Washington University School of Medicine